CLINICAL TRIAL: NCT04210856
Title: Effects of Landscapes on the Brain: Assessment of Neurophysiological Response in Healthy and Depressed Individuals to Different Landscape Quality Exposures in Singapore
Brief Title: Effects of Landscapes on the Brain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: National University Hospital, Singapore (Other); National Parks Board, Singapore (Other); Ministry of National Development, Singapore (Other Government)
Responsible Party: Principal Investigator, Agnieszka Olszewska-Guizzo, Principal Investigator, National University of Singapore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: R-722-000-010-490
Record Dates: First submitted 2019-12-19; First posted 2019-12-26 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Depression; Stress; Anxiety Disorders
Keywords: landscape; exposure; EEG; fNIRS; depression; stress; urban; anxiety; contemplative
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: non-randomised within subjects clinical trial.
Masking Description: participants do not know the hypothesis of a study, other people cannot influence the brainwave reaction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sequence of Landscape exposures (Experimental): All participants undergo the procedure of visiting all landscape exposures in a random order.
  Interventions: Other: Contemplative landscape exposure

INTERVENTIONS:
Other: Contemplative landscape exposure — landscapes classified as contemplative (through a CLM psychometric measure) are expected to elicit different brainwave oscillations as compared to non-contemplative ones.

SUMMARY:
There is an established consensus between researchers that the contact with natural environments has beneficial influence on mental health and well-being of people exposed to them. The knowledge in this area is based mostly on the correlational analyses, but more research is needed to explore the causal relationships between the human and his environment. More specifically, in order to identify specific restorative mechanisms in response to the specific types and components of the designed landscapes, especially in the highly urbanized context.

This study will attempt to find the psychophysiological responses in human brain to landscapes videos (in the lab), and real landscapes with different visual quality, carefully pre-selected and analysed in terms of landscape composition. In the study the rigorous experimental protocol will be administered in order to acquire qualitative and quantitative data both self-reported and measured by neuroscience tools, in order to demonstrate the causal effect of landscape exposure on the brain activity patterns and mood of healthy and depressed individuals.

DETAILED DESCRIPTION:
Understanding of the impact of urban green landscapes with different design and levels of contemplativeness on brain function may pave the way to more scientifically informed and more healthy planning and design of urban living environment.

Also the exposure to certain types of landscapes may be useful in mental health promotion and support for the existing treatments in patients with depression.

Specific aims The aim of the study is to assess the effects of passive exposure (viewing) images of differently designed landscapes on the brain activity of two groups: 1) healthy individuals and 2) patients with depression, using electroencephalography (EEG) and Functional Near-Infrared Spectroscopy (fNIRS). The investigators also want to compare effects of exposure to images with the in-situ immersion with the real environment.

Following the assumption that there are certain types and components of the living environments that influence our mental health and well-being even if one is passively exposed to them, the investigators want to to assess the effects of passive exposure to three differently designed, representative landscapes on the brain activity of healthy individuals. And to compare effects of exposure to images with the in-situ immersion with the real environment.

Hypothesis The investigators hypothesise that landscapes, that the Therapeutic Garden, which also achieved a high score in the Contemplative Landscape expert evaluation scale, will induce the brain activity patterns commonly associated with the relaxation, and bottom-up attention, unlike the other selected sites with lower scores. Additionally, the investigators hypothesize that in the real landscape exposures they will observe this phenomenon more intensely than in the case of images exposure.

PARTICIPANTS The investigators will recruit 100 right-handed healthy participants aged 21-75 y.o. Based on previous studies using fNIRS to study motor task (Siedel et al., 2017), the minimum number of participants is 50 participants per group. As a result, recruitment of 100 participants in order to ensure the minimal number of participants in the case of dropouts was proposed.

Exclusion criteria:

* Left-handedness;
* serious visual impairment; reported psychiatric, neurological or cognitive diseases;
* reported use of medication that could alter the functioning of the Central Nervous System at the time of the experiment;
* existence of a pacemaker, intracranial electrodes, implanted defibrillator or plates,
* otologic surgery in the last 12 months.

The investigators will also recruit 100 right-handed patients with diagnosed depression at the Neuroscience Clinic or Psychiatric ward in National University Hospital (NUH)

Inclusion criteria:

* Age of 21 to 75
* Right-handed only
* They must suffer from depressive disorder,

Exclusion criteria:

* Major neurological disorders e.g. epilepsy, stroke
* Any form of cancer
* Major heart diseases: e.g. ischemic heart disease
* Major lung diseases: e.g. chronic obstructive pulmonary disorder.
* Major liver disease e.g. liver failure
* Major kidney disease e.g. kidney failure.

Recruitment:

The target individuals will be recruited by word of mouth. The principal investigator or co-investigator will approach the participants who fulfil the inclusion criteria and explain the purpose and procedure of this project. If the participant agrees to participate in this project, he or she will sign the consent form after reading the Participant Information Sheet that provides information about this study. Then the investigators will arrange the time schedule to perform the sessions for the participant.

Ethics approvals:

For healthy participants: Ref #: S-18-352 For patients: NHG DSRB Ref # 2018/01036

METHODS NEUROIMAGING EQUIPMENT The NIRS and EEG data will be collected using NIRSport (LLC NIRx Medical Technologies). The former consists of 8 illumination sources and 8 detection sensors with two wavelengths of 760nm & 850nm, yields 128 data channels, with a sampling rate 62.5 Hz.

The latter is V-Amp 16-channel portable EEG system, with active -dry type of electrodes (actiCAP Xpress), bandwidth of 0Hz (DC) - 500Hz(-3 dB) and sampling rate up to 20.000 Hz. Both devices are lightweight, portable and adjusted to the outdoor environment data collection, and mountable on one single cap to reduce discomforts of long data collection for participants.

EXPERIMENTAL DESIGN

This study is a non-randomised within subjects clinical trial. All participants will attend four landscape viewing sessions while having their brains imaged using the fNIRS and EEG (both machines combined into 1 cap), they will also complete an emotional state assessment questionnaire (Profile of Mood States - POMS, [Shacham,1983]), landscape preference questionnaire (Self-Assessment Manikin) and Beck Depression Inventory (BDI).The latter will serve as a control for the extreme scores in the healthy population i.e. if a healthy patricipants score shows that this participant may suffer from undiagnosed depression their data may be eliminated from the further analysis. The participant with high depression score will be advised to seek clinical assessment by psychiatrist. First session will take place in the research room at the BIGHEART premises (lab indoor environment), and three remaining sessions in the 3 oudoor preselected sites (real landscapes) - see Table 1.

Table 1. Location of the data collection sessions, and estimated time of participation Viewing session Site Adress Estimated Time

1. Lab (indoors) BIGHEART, 14 Medical Drive, #14-01. 50min
2. Site 01 (outdoors) Therapeutic Garden @Hortpark, 33 Hyderabad Rd, Singapore 20min
3. Site 02 (outdoors) Casa Clementi, Clementi Ave 1, Singapore 20min
4. Site 03 (outdoors) Sheltered sidewalk, 32 New Market Rd, Singapore 20min

Indoor Experimental protocol The first, lab-based session will start with informed consent, and completion of pre-experiment POMS (profile of mood state) questionnaire. The participant code will be then attributed to each participant, their personal information will not be used any more in the study: they will not be needed in the future and will not need to be stored. All electronic devices in the room are to be switched off except necessary data collection equipment. The room temperature and humidity will be kept the same across all participants and conditions. Before the data collection each participant will have the multimodal NIRS and EEG device positioned on their heads.

Participants will be instructed to sit comfortably on a chair and without talking or moving calmly observe the landscape views displayed in front of them, while simultaneously their brain signals will be recorded using NIRS and EEG. Resting state activity for each participant will be recorded preceding the display of the videos.

There will be 1 minute of resting state (baseline) recording followed by the landscape 9 fixed-frame videos viewing, displayed for 20 seconds, repeated 3 times each in a randomized order to avoid order bias. In between the landscapes there will be a fixation cross displayed for 5 seconds. So the overall time of recording EEG/fNIRS signal will take about 13 minutes.

After that four questionnaires will be completed by the participant, including respectively: (1) post-experimental POMS questionnaire, (2) landscape preference questionnaire, (3) Depression scale (BDI questionnaire) and (4) socio-demographic questionnaire. There are some questions that may be deemed sensitive to some participants, in this case they are allowed to skip an uncomfortable question.

The whole procedure (including explanation, consent taking, questionnaire and cognitive tasks) should be completed within 50 min. The fNIRS and EEG signals recorded during landscapes viewing as well as each cognitive task will be stored in the computer.

Outdoor Landscape Experiment multimodal NIRS and EEG In this study participants will be invited to the site session, morning (between 10AM and 12PM) or afternoon (between 2PM and 4PM). For the safety of participants and sound quality of the study design the weather during the session must be normalized: not too hot, dry with clear or partly cloudy sky. In the event of the bad weather conditions (rain, storm, heat wave) the sessions will be postponed. The travel expenses for a participant getting to the sites will be included in the reimbursement.

Because of possibility of disruption of the public space (especially in the case of Site 03), only up to 2 participants can have the session scheduled at the same time.

After completing the pre-experimental POMS questionnaire, participants will be seated in front of an actual landscape view, and advised to calmly observe it, without moving. The researchers will control for the outdoor brightness using the standard light-meter, thus the onsite data collection should be performed at the similar time of a day, with the similar weather conditions and keeping all other factors (such as other visitors and any other distracting phenomena) at the similar levels across all participants.

All the rest of the outdoors experimental procedures will be similar to the laboratory procedure except no consent (the consent signing will take place prior to the outdoors sessions), no socio-demographic and no BDI questionnaire will be performed. Participants will be seated in front of each of 3 landscape views at a location, and for the baseline recording the white glasses will be put on their eyes to cover the view. After baseline recording they will passively watch the landscape view for 1 minutes.

After data collection the devices will be dismounted from the head of participant and the POMS questionnaire will be performed.

The time of the participation in the outdoor session will be therefore shorter, estimated at 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age of 21 to 75
* Right-handed only
* (They must suffer from depressive disorder)

Exclusion Criteria:

* Major neurological disorders e.g. epilepsy, stroke
* Any form of cancer
* Major heart diseases: e.g. ischemic heart disease
* Major lung diseases: e.g. chronic obstructive pulmonary disorder.
* Major liver disease e.g. liver failure
* Major kidney disease e.g. kidney failure.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2021-07-09 (Actual)

PRIMARY OUTCOMES:
EEG power in alpha band | 5 minutes
  predictor of positive affect and positive mental health outcomes, measured with EEG
EEG power in beta band | 5 minutes
  more beta in the right temporal lobes associated with stimuli-driven attention, measured with EEG
fNIRS haemodynamics | 5 minutes
  decreased oxy-hemoglobin in the frontal part of the brain indicates more relaxation

SECONDARY OUTCOMES:
Profile of mood states | 30 minutes
  self-reported, pre-and post- stimulation Profile of Mood States (POMS) scale measures the change in the momentary mood, giving as an outcome measure the Total Mood Disturbance (TMD), where 1 is neutral, and above 1 is disturbed mood.
landscape preference measured with self-assessment manikin scale. | 30 minutes
  measured using pictorial Self-Asessment Manikin (SAM) where score ranged from -3 to +3, where the lower the score the less positive (valence + arousal) emotions are caused by looking at the view

CONTACTS AND LOCATIONS:
Overall Officials: Ho Roger, MDD, Principal Investigator — NUHS
Locations (1):
- Institute for Health Innovation & Technology (iHealthtech), Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No